CLINICAL TRIAL: NCT00662103
Title: Comparison of Aerobic and Resistance Exercise in Older Breast Cancer Survivors
Brief Title: Aerobic Exercise, Resistance Exercise, or Flexibility and Relaxation Training in Inactive Older Female Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CDR0000593410; R01CA120123 (NIH); P30CA069533 (NIH); OHSU-CR00005268; OHSU-IRB00003316; NCT00665080 (obsolete NCT alias)
Record Dates: First submitted 2008-04-18; First posted 2008-04-21 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer; Cancer Survivor; Fatigue; Long-term Effects Secondary to Cancer Therapy in Adults; Psychosocial Effects of Cancer and Its Treatment
Keywords: fatigue; long-term effects secondary to cancer therapy in adults; psychosocial effects of cancer and its treatment; cancer survivor; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Breast Carcinoma In Situ | interventions — Therapeutics; Psychiatric Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- progressive, aerobic exercise program (Active Comparator): Patients undergo aerobic exercise training over approximately 45 minutes (not including warm-up or cool-down exercises) 3 days a week for 18 months.
  Interventions: Behavioral: exercise intervention; Other: laboratory biomarker analysis; Other: questionnaire administration; Other: survey administration; Procedure: assessment of therapy complications; Procedure: fatigue assessment and management; Procedure: management of therapy complications; Procedure: psychosocial assessment and care
- progressive, resistance exercise program (Active Comparator): Patients undergo resistance exercise training 3 days a week for 18 months.
  Interventions: Behavioral: exercise intervention; Other: laboratory biomarker analysis; Other: questionnaire administration; Other: survey administration; Procedure: assessment of therapy complications; Procedure: fatigue assessment and management; Procedure: management of therapy complications; Procedure: psychosocial assessment and care
- flexibility and relaxation training [control] (Active Comparator): Patients perform a series of whole body flexibility (stretching) and relaxation (guided imagery, progressive neuromuscular relaxation, focused breathing) exercises 3 days a week for 18 months.
  Interventions: Other: laboratory biomarker analysis; Other: questionnaire administration; Other: survey administration; Procedure: assessment of therapy complications; Procedure: fatigue assessment and management; Procedure: management of therapy complications; Procedure: psychosocial assessment and care

INTERVENTIONS:
Behavioral: exercise intervention — Arm I (progressive, aerobic exercise program): Patients undergo aerobic exercise training over approximately 45 minutes (not including warm-up or cool-down exercises) 3 days a week for 18 months.
  Arm II (progressive, resistance exercise program): Patients undergo resistance exercise training 3 days a week for 18 months.
  Arms: progressive, aerobic exercise program; progressive, resistance exercise program
Other: laboratory biomarker analysis — All biomarkers will be measured from urine, blood and plasma obtained from participants by the Oregon Health & Science University (OHSU) General Clinical Research Center (GCRC). Upon exit from the study we will confirm the presence/absence of metastatic disease, via verbal verification by the subject, in order to ensure that biomarkers were primarily reflective of bone turnover changes and not to metastases.
Other: questionnaire administration — Patients complete questionnaires at baseline and periodically during the study to assess demographic (i.e., age, income) and disease-specific (i.e., stage, treatment) variables, self-report mental and physical function, presence of chronic medical conditions, symptoms, fatigue, exercise outside the study exercise intervention, dietary intake, and psychosocial function.
Other: survey administration — Administered at measured at baseline, 3, 6, 12, and 18 months
Procedure: assessment of therapy complications — Follow-up every 6 months (measured at baseline, 3, 6, 12, and 18 months )
Procedure: fatigue assessment and management — The Schwartz Cancer Fatigue (SCF) scale, a 6-item scale that specifically assesses the level of subjective fatigue that the participant is currently experiencing. The SCF has been used to measure fatigue in previous exercise studies. The Piper Fatigue Scale (PFS) consists of 22 items and four subscales: behavioral/severity, affective meaning, sensory and cognitive/mood. The scale has been shown to detect reductions in fatigue in cancer patients undergoing behavioral interventions to reduce fatigue, including exercise. Responses are averaged for subscale and total scores with higher scores indicating more fatigue. The PFS has been used to measure fatigue in previous studies of illness and/or medical treatments. 15 minute survey
Procedure: management of therapy complications — An interim safety/efficacy review will occur after the first half of enrolled participants completes their 3 month testing appointment (or after 3 months of exercise). The interim safety review will be overseen by OHSU NCI-designated Cancer Institute, while the efficacy review will be conducted by an independent monitor, Dr. George Knafl, a biostatistician in the OHSU School of Nursing, who is not a member of the study personnel.
Procedure: psychosocial assessment and care — We will include a 6-item measure of self-efficacy for exercise that has been validated in adults (Nigg, 2002) and has been used by Dr. Bennett (Co-I) in current work in cancer survivors. 5 min. survey

SUMMARY:
RATIONALE: Aerobic exercise, resistance exercise, and flexibility and relaxation training may reduce fatigue and improve the health and quality of life of breast cancer survivors. It is not yet known which type of exercise is more effective for inactive older female breast cancer survivors.

PURPOSE: This randomized clinical trial is studying aerobic exercise to see how well it works compared with resistance exercise or flexibility and relaxation training in improving the health and quality of life of inactive older female breast cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary:

* Compare the effects of aerobic exercise vs flexibility and relaxation training (control) on fatigue, aerobic capacity, functioning, and health outcomes in inactive older female breast cancer survivors.
* Compare the effects of resistance exercise vs flexibility and relaxation training (control) on fatigue, muscle strength, functioning, and health outcomes.

Secondary:

* Compare the relative effects of aerobic exercise vs resistance exercise on fatigue, physical functioning, physical health, and mental health.
* Determine the mediating effects of fatigue and fitness on the relationship between exercise and physical functioning.
* Compare the individual and relative effects of aerobic exercise vs resistance exercise vs flexibility and relaxation training (control) on body composition and on biomarkers of cancer recurrence.

OUTLINE: Patients are stratified according to current use of hormone manipulation therapy (none vs tamoxifen vs arimidex). Patients are randomized to 1 of 3 intervention arms.

* Arm I (progressive, aerobic exercise program): Patients undergo aerobic exercise training over approximately 45 minutes (not including warm-up or cool-down exercises) 3 days a week for 18 months. During the first 12 months, patients attend supervised aerobic exercise sessions 2 days a week and complete 1 home-based aerobic exercise session using a modified exercise program designed by the investigative team. During the final 6 months, patients undergo aerobic exercise using an at-home program designed by the investigative team. Aerobic exercise training comprises simple stepping routines using benches of various heights while wearing a wrist monitor to record heart rate. Volume of aerobic exercise, determined by intensity (heart rate at percentage of heart rate reserve tailored to the patient) and duration (minutes in the target heart rate range), is gradually and progressively increased over the first 9 months of the exercise program. Exercise volume remains at a moderate level for the remainder of the program to provide an optimal physiologic challenge at a safe and tolerable level.
* Arm II (progressive, resistance exercise program): Patients undergo resistance exercise training 3 days a week for 18 months. During the first 12 months, patients attend supervised resistance exercise sessions 2 days a week and complete 1 home-based resistance exercise session using a modified exercise program designed by the investigative team. During the final 6 months, patients undergo resistance exercise using an at-home program designed by the investigative team. Resistance exercise training comprises the use of hand weights and barbells (for upper body resistance) and exercises in weighted vests (for lower body resistance). Patients wear a weighted vest while performing lower body strength training (chair rises, 90-degree squats, toe raises, forward lunges, lateral lunges). Patients use hand weights for upper body strength training (upright row, 1-arm row, overhead press, chest press, chest fly, biceps curl, triceps extension). Volume of strength training, determined by intensity (weight tailored to the patient) and duration (number of sets), is gradually increased from low weight and high number of repetitions to more weight and fewer repetitions over the first 6 months of the training period. Exercise volume remains at a moderate intensity for the remainder of the training period to provide an optimal physiologic challenge at a safe and tolerable level.
* Arm III (flexibility and relaxation training [control]): Patients perform a series of whole body flexibility (stretching) and relaxation (guided imagery, progressive neuromuscular relaxation, focused breathing) exercises 3 days a week for 18 months. During the first 12 months, patients attend supervised flexibility and relaxation exercise sessions 2 days a week and complete 1 home-based flexibility and relaxation exercise session using a modified exercise program designed by the investigative team. During the final 6 months, patients undergo flexibility and relaxation exercises using an at-home program designed by the investigative team.

Muscle strength (measured by a one-repetition maximum test), aerobic capacity (measured by a 6-minute walk test), functional arm strength (measured by grip dynamometer), physical functioning (measured by the Physical Performance Battery), flexibility (measured by the Chair Sit and Reach Test and the Back Scratch Test), balance (measured by a one-legged stance [Romberg] test and a timed stance test), lymphedema (measured by the circumference of the upper arm, wrist, and a finger), body composition (measured by dual energy x-ray absorptiometry), and bone mineral density of the heel (measured by ultrasound) are assessed at baseline and periodically during the study. Patients also undergo blood and urine sample collection for cancer recurrence biomarker and bone remodeling biomarker studies.

Patients complete questionnaires at baseline and periodically during the study to assess demographic (i.e., age, income) and disease-specific (i.e., stage, treatment) variables, self-report mental and physical function, presence of chronic medical conditions, symptoms, fatigue, exercise outside the study exercise intervention, dietary intake, and psychosocial function.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer

  * Stage 0-III disease
* Completed chemotherapy or radiotherapy > 2 years ago
* Is not a regular participant in moderate aerobic exercise (i.e., jogging, swimming) or moderate resistance exercise (> 3 times/week for ≥ 30 minutes/session) OR in vigorous aerobic or resistance exercise (> 3 times/week for ≥ 20 minutes/session)
* No stage IV breast cancer
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Has obtained medical clearance to participate in study exercise programs
* No cognitive difficulties that would preclude answering the survey questions, participating in the performance tests, or giving informed consent
* No medical condition or movement or neurological disorder that would contraindicate participation in moderate intensity exercise training, as determined by physician clearance and the Principal Investigator

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent medication that would contraindicate participation in moderate intensity exercise training, as determined by physician clearance and the Principal Investigator
* Concurrent hormonal therapy (e.g., selective estrogen receptor modulator (SERM) or aromatase inhibitor) for breast cancer allowed

Ages: 65 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 115 (Actual)
Dates: Start 2008-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Comparison of the effects of aerobic exercise vs flexibility and relaxation training (control) on fatigue, aerobic capacity, functioning, and health outcomes as measured at baseline and at 3, 6, 12, and 18 months | baseline,3 ,6 ,12, and 18 months
Comparison of the effects of resistance exercise vs flexibility and relaxation training (control) on fatigue, muscle strength, functioning, and health outcomes as measured at baseline and at 3, 6, 12, and 18 months | baseline, 3 , 6 ,12, and 18 months

SECONDARY OUTCOMES:
Comparison of the relative effects of aerobic exercise vs resistance exercise on fatigue, physical functioning, physical health, and mental health as measured at baseline and at 3, 6, 12, and 18 months | baseline, 3, 6, 12, and 18 months
Determination of the mediating effects of fatigue and fitness on the relationship between exercise and physical functioning as measured at baseline and at 3, 6, 12, and 18 months | baseline, 3, 6, 12, and 18 months
Comparison of the individual and relative effects of aerobic exercise vs resistance exercise vs flexibility and relaxation training (control) on body composition and on biomarkers of cancer recurrence as measured at baseline and at 3, 6, 12, and 18 ... | baseline, 3, 6, 12, and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Winters-Stone, PhD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Winters-Stone KM, Torgrimson-Ojerio B, Dieckmann NF, Stoyles S, Mitri Z, Luoh SW. A randomized-controlled trial comparing supervised aerobic training to resistance training followed by unsupervised exercise on physical functioning in older breast cancer survivors. J Geriatr Oncol. 2022 Mar;13(2):152-160. doi: 10.1016/j.jgo.2021.08.003. Epub 2021 Aug 21. PMID 34426142
- [Derived] Winters-Stone KM, Wood LJ, Stoyles S, Dieckmann NF. The Effects of Resistance Exercise on Biomarkers of Breast Cancer Prognosis: A Pooled Analysis of Three Randomized Trials. Cancer Epidemiol Biomarkers Prev. 2018 Feb;27(2):146-153. doi: 10.1158/1055-9965.EPI-17-0766. Epub 2017 Nov 15. PMID 29141853